CLINICAL TRIAL: NCT04600570
Title: Ultrasonographic Measurement of the Optic Nerve Sheath Diameter in the Taiwanese Healthy Volunteers and Its Associating Factors
Brief Title: Ultrasonographic Measurement of the Optic Nerve Sheath Diameter in the Taiwanese Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202008032RINC
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Normal Diameter of Optic Nerve
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: ultrasound — ultrasound measurement for optic nerve outer diameter

SUMMARY:
The investigators aimed to analyze the ONSD diameters and its associated factors in Taiwanese healthy volunteers. We plan to recruit 150 healthy volunteers aged more than 20 years old. The ONSD and its associated factors will be measured and recorded by ultrasound from September 2020 to August 2021.

DETAILED DESCRIPTION:
Ultrasound measurement of optic nerve sheath diameter (ONSD) had been considered as a non-invasive way to distinguish the presence of elevated intracranial pressure (ICP). Besides detecting elevated ICP in various neurological diseases, ONSD can also be applied to cardiac arrest survivors as one of the prognostic factors. It is a simple, quick, repeatable technique without the need of contrast medians. In order to make precise interpretations, the database of the normal distribution of ONSD and its associated factors in healthy volunteers is necessary. The majority of previous reports are from Western countries, and limited reports of ONSD in the Asian population have high variability.

Therefore, collecting local data of ONSD in Taiwan is important. In this study, the investigators aimed to analyze the ONSD diameters and its associated factors in Taiwanese healthy volunteers. The investigators planed to recruit 150 healthy volunteers aged more than 20 years old. The ONSD and its associated factors will be measured and recorded by ultrasound from September 2020 to August 2021.

ELIGIBILITY:
Inclusion Criteria:

adult volunteer aged more than 20 years

Exclusion Criteria:

aged less than 20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
optic nerve outer diameter | 60 days
  optic nerve outer diameter

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — NTUH
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No